CLINICAL TRIAL: NCT05641103
Title: PREDIGA 2: Spanish Acronym of "Educational and Diagnostic Project for Gaucher and ASMD"
Acronym: PREDIGA-2
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: PREDIGA-2
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-05

CONDITIONS: Gaucher Disease; Acid SphingoMyelinase Deficiency; ASMD; Niemann-Pick Diseases; Splenomegaly
MeSH Terms: conditions — Gaucher Disease; Niemann-Pick Diseases; Splenomegaly | interventions — Splenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patient with splenomegaly or splenectomy — No interventional study

SUMMARY:
The study of splenomegaly, and the follow-up of splenectomized patients, is one of the causes of referral of these patients to pediatric gastroenterology and oncohematology clinics, and adult internal medicine and hematology. It has been described that 0.3% of hospital admissions is for this reason.

The study and management of splenomegaly is well described among the different medical specialties to which these patients arrive. After the application of the different algorithms and the different studies that are carried out, these splenomegaly are identified as being of hepatic, infectious, inflammatory, congestive, hematological origin and primary causes. Despite these studies of splenomegaly, approximately 10-15% of these patients still remain undiagnosed.

The objective of the present study is to increase the diagnostic sensitivity of these unknown splenomegalys, or unknown splenomegaly patients who remain in consultations, using the usual diagnostic clinical procedures of unknown splenomegaly and unknown splenectomy patients, where the investigators include the extraction of a blood sample for dry drop test (DBS), where the determination of the enzymatic/genetic activity will be carried out for Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD) , analysis of LisoGl1 and LisoSM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes.
* Patients who present signs, assessed instrumentally or with laboratory tests, of unknown splenomegaly, defined as a palpable spleen ≥ 1cm from the costal margin or diagnosed by ultrasound, magnetic resonance imaging (MRI) or computed tomography (CT) of the spleen.
* Splenectomy patient with no diagnosis of the origin of the splenomegaly of unknown origin.
* Patients with splenomegaly or splenectomy without diagnosis but identified with ITP (Idiopathic Thrombocytopenic Purpura)
* Patient who gives his consent to participate in the study.

Exclusion Criteria:

* Splenomegaly due to portal hypertension (documented by abdominal ultrasound or other instrumental test) due to liver disease
* Hematologic malignancy [documented by positive physical exam + blood smear or fine needle aspiration (FNA) or bone marrow biopsy]
* Hemolytic anemia and/or thalassemia
* Patients who cannot meet the requirements of the protocol due to mental and/or cognitive alterations, uncooperative patients, educational limitations and understanding of written language
* Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with splenomegaly and unknown splenectomized
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD) | 36 months
  Determinate the prevalence of Gaucher disease (GD) and acid sphingomyelinase deficiency (ASMD)

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital de Poniente, El Ejido, Almería
  - Hospital Universitario de Badajoz, Badajoz, Badajoz
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario Juan Ramón Jiménez, Huelva, Huelva
  - Complejo Hospitalario Universitario La Coruña - CHUAC, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago - CHUS, Santiago de Compostela, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias - HUCA, Oviedo, Principality of Asturias
  - CAU Salamanca, Salamanca, Salamanca
  - Hospital Universitario Joan XXIII, Tarragona, Tarragona
  - Hospital Universitario de Galdácano, Galdakao, Vizcaya

IPD SHARING:
Plan to Share IPD: No